CLINICAL TRIAL: NCT07045194
Title: A Prospective, Multi-center, Single-blind, Randomized (1:1), Non-inferiority Study Comparing Clinical Outcomes of the Virtue® Sirolimus AngioInfusion™ Balloon (SAB) to the AGENT™ Paclitaxel Drug-Coated Balloon (DCB) in the Treatment of Coronary Artery In-stent Restenosis (ISR).
Brief Title: Virtue® SAB in the Treatment of Coronary ISR Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orchestra BioMed, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol - 0072
Record Dates: First submitted 2025-06-16; First posted 2025-07-01 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Coronary Artery Disease
Keywords: In-Stent Restenosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Virtue SAB (Experimental): Coronary PCI, Sirolimus AngioInfusion Balloon (SAB)
  Interventions: Device: Virtue Sirolimus AngioInfusion Balloon
- AGENT™ DCB (Active Comparator): Coronary Angioplasty, AGENT™ Paclitaxel Drug-Coated Balloon (DCB)
  Interventions: Device: AGENT™ Paclitaxel Drug-Coated Balloon

INTERVENTIONS:
Device: Virtue Sirolimus AngioInfusion Balloon — Percutaneous Coronary Intervention
  Arms: Virtue SAB
Device: AGENT™ Paclitaxel Drug-Coated Balloon — Percutaneous Coronary Intervention
  Arms: AGENT™ DCB

SUMMARY:
A prospective, multi-center, single-blind, randomized (1:1), non-inferiority study comparing clinical outcomes of the Virtue® Sirolimus AngioInfusion™ Balloon (SAB) to the AGENT™ Paclitaxel Drug-Coated Balloon (DCB) in the treatment of coronary artery in-stent restenosis (ISR).

DETAILED DESCRIPTION:
The Virtue® ISR trial is a prospective, multi-center, single-blind, randomized (1:1), non-inferiority study. The Virtue® Sirolimus AngioInfusion™ Balloon (SAB) will be compared to the AGENT Paclitaxel Drug-Coated Balloon (DCB) in the treatment of coronary artery in-stent restenosis (ISR).

ELIGIBILITY:
Inclusion Criteria:

* In-stent restenosis (one or two stent layers) in a lesion previously treated with drug- eluting (DES) or bare metal stents (BMS) in a native coronary artery.
* The target lesion is in a vessel with a reference vessel diameter ≥ 2.0 mm and ≤ 4.0 mm by visual assessment.
* The subject has only one critical ISR lesion.
* The subject may have one other critical lesion in a non-target vessel that must be treated before the Target Lesion (TL).
* Target lesion length must be ≤ 26 mm and must be completely coverable by only one Virtue® or AGENT™ balloon. The balloon can extend up to 5 mm proximal or distal beyond the edge of the target stented length.
* The target lesion must have one of the following:
* Visually estimated stenosis of ≥ 70% and <100% diameter stenosis, OR
* Visually estimated stenosis ≥ 50% and < 70% with one of the following:
* abnormal fractional flow reserve (FFR) including Angio based FFR ≤ 0.80, or;
* abnormal instantaneous wave-free ratio (iFR) or resting full-cycle ratio (RFR) ≤ 0.89, or;
* abnormal stress or imaging stress test, or;
* ischemic symptoms referable to the target lesion
* Involved in a NSTEMI or Acute Coronary Syndrome (ACS) event with decreasing enzymes
* Target lesion must be successfully pre-treated according to standard of care with an achieved residual stenosis of ≤ 30% by visual estimate with TIMI grade flow of 3 prior to randomization.

Exclusion Criteria:

* Subject has a left ventricular ejection fraction < 30% within 6 months.
* Subject was treated by PCI or another coronary intervention within the last 30 days.
* Planned PCI or CABG after the index procedure.
* Subjects with STEMI < 72 hours prior to index procedure and those with NSTEMI who have increasing biomarkers within 12 hours of the index procedure.
* If single-layer ISR, any previous treatment (other than balloon angioplasty alone) of the target vessel for restenosis. If double-layer ISR, any treatment (other than balloon angioplasty alone) of the double-layer ISR restenosis.
* Target lesion is located within a saphenous vein graft or an arterial graft.
* Thrombus is present in the target vessel.
* > 50% stenosis of an additional lesion proximal or clinically significant distal (>2.0mm RVD) to the target lesion.
* A dissection in the target lesion requiring treatment with a stent post pre-dilatation.
* The target ISR lesion has more than two layers of previously placed stents.
* Subject has critical unprotected left main coronary artery disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) at 12 months | 12 months
  Defined as a composite of cardiac death (CD), non-fatal target vessel myocardial infarction (MI) SCAI definition, and ischema-driven target lesion revascularization (TLR)

SECONDARY OUTCOMES:
Target Lesion Failure (TLF) Comparison at 12 months | 12 months
  Target Lesion Failure (TLF) at 12 months of subjects treated with Virtue® SAB compared to a PBA Performance Goal.

CONTACTS AND LOCATIONS:
Overall Officials: Dean Kereiakes, MD, Principal Investigator — Lindner Center for Research at Christ Hospital; Allen Jeremias, MD, Principal Investigator — St. Francis Hospital & Heart Center
Locations (2):
- United States (2):
  - St. Francis Hospital, Roslyn, New York
  - The Lindner Center for Research at Christ Hospital, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No